CLINICAL TRIAL: NCT01107717
Title: Durability of Early Initial Combination Therapy With Exenatide/Pioglitazone/Metformin vs Conventional Therapy in New Onset Type 2 Diabetes
Brief Title: Durability of Combination Therapy With Exenatide/Pioglitazone/Metformin vs. Conventional Therapy in New Onset T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American Diabetes Association (Other); Amylin Pharmaceuticals, LLC. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20080456H; 5R01DK103841-03 (NIH)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Diabetes
Keywords: type 2 diabetes; new onset; combination therapy; new onset type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin; Glyburide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple Therapy (Experimental): initiation a combination of metformin (1000 mg), pioglitazone (15 mg) and exenatide (5 microgram bid) at the time diabetes is diagnosed
  Interventions: Drug: metformin\pioglitazone\exenatide
- conventional therapy (Active Comparator): sequential addition of metformin, glyburide and basal insulin
  Interventions: Drug: metformin, glyburide and glargine

INTERVENTIONS:
Drug: metformin\pioglitazone\exenatide — metformin (1000 mg), pioglitazone (15 mg) and exenatide (5 microgram bid) are started and dose is up titrated to achieve HbA1c < 6.5%
  Arms: Triple Therapy
Drug: metformin, glyburide and glargine — subjects are started on metformin 500 mg bid and dose is up titrated and glyburide (up to 5 mg) and glargine are sequentially added to maintain HbA1c < 6.5%
  Arms: conventional therapy

SUMMARY:
Type 2 diabetes is a systemic metabolic disease with significant morbidity and mortality due to damaging blood vessels. Increased blood sugar level is a hallmark of diabetes and is an contributes to the development of many of its complications. Multiple defects, e.g. impaired insulin secretion and impaired insulin action, contribute to the development of the disease. The aim of this study is to test the efficacy and durability of combination of drugs which correct the defects that lead to the development of diabetes on achieving adequate and durable control of blood sugar levels. Achieving adequate and durable control of blood sugar will prevent many of diabetes complications.

DETAILED DESCRIPTION:
Subjects will be randomized (using a table of random numbers) to receive, in open label fashion, one of the following treatment regimens: (i) Group I will be started on pioglitazone (15 mg/day) plus metformin (1000 mg/day) with the supper meal and exenatide (5 mcg s.c. bid 30 min before breakfast and supper) and up-titrated to 45 pioglitazone plus 2000 metformin and 10 mcg s.c. bid exenatide to achieve HbA1c <6.0%; (II) Group II will be started on metformin, 1000 mg with breakfast and 1000 mg with supper, glyburide and basal insulin will be added and up titrated to achieve HbA1c <6.0% The study team will compare the efficacy of two therapeutic regimens: (i) triple therapy (pioglitazone, metformin, exenatide) at the time of diagnosis of T2DM versus (ii) stepwise therapy starting with metformin and subsequent addition of sulfonylurea and basal insulin (i.e., the "standard" approach) in achieving this goal. The first intervention is based on the novel concept of initiating therapy at the time of diagnosis with combination therapy using agents that correct specific pathophysiologic defects that are characteristic of T2DM (insulin resistance and beta cell failure). The second intervention is based upon stepwise addition of antidiabetic agents to reduce the HbA1C according to the current ADA therapeutic recommendation.

ELIGIBILITY:
Inclusion Criteria:

* subjects with type 2 diabetes diagnosed during the past 2 years,
* above 18 years of age,
* drug naive, or have been on metformin less than 3 months

Exclusion Criteria:

* subjects with type 1 diabetes or GAD positive subjects or subjects with long standing diabetes (>2 years) or subjects who are not drug naive or have been on metformin more than 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2009-01; Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Texas Diabetes Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with local investigators
Supporting Information: Study Protocol, SAP
Time Frame: At study completion after publication in a peer review journal

REFERENCES:
- [Result] Abdul-Ghani M, Puckett C, Adams J, Khattab A, Baskoy G, Cersosimo E, Triplitt C, DeFronzo RA. Durability of Triple Combination Therapy Versus Stepwise Addition Therapy in Patients With New-Onset T2DM: 3-Year Follow-up of EDICT. Diabetes Care. 2021 Feb;44(2):433-439. doi: 10.2337/dc20-0978. Epub 2020 Dec 3. PMID 33273042
- [Derived] Abdul-Ghani M, Puckett C, Abdelgani S, Merovci A, Lavrynenko O, Adams J, Triplitt C, DeFronzo RA. Glycemic and non-glycemic benefits of initial triple therapy versus sequential add-on therapy in patients with new-onset diabetes: results from the EDICT study. BMJ Open Diabetes Res Care. 2025 Apr 27;13(2):e004981. doi: 10.1136/bmjdrc-2025-004981. PMID 40288809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Newly diagnosed T2DM participants
Period: Overall Study
Arm/Group | Triple Therapy | Conventional Therapy
Started | 157 | 161
Completed | 103 | 114
Not Completed | 54 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 103 | 114 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (1) | 47 (1) | 45.5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 72 | 124
  Male | 51 | 42 | 93
Race/Ethnicity, Customized [Number; unit: participants]
  Mexican Americans | 73 | 75 | 148
  Caucasian | 15 | 15 | 30
  Other | 15 | 24 | 39
Region of Enrollment [Number; unit: participants]
  United States | 103 | 114 | 217
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dl] | 203 (6) | 200 (6) | 201.5 (6)
Diabetes Duration at start [Mean (Standard Deviation); unit: Months] | 4.8 (0.5) | 5.2 (0.5) | 5 (0.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.4 (1.1) | 36.1 (1.1) | 36.25 (1.1)
Baseline HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — percentage of Hba1c.
  percentage of glycated hemoglobin | 9.0 (0.2) | 8.8 (0.2) | 8.9 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Level
Description: subjects will be followed for 3 years and the HbA1c measured at this time to provide the values for each arm as defined for the primary outcome of the study
Time Frame: at the end of the study (3 years)
Measure: Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Triple Therapy | Conventional Therapy
Number analyzed (Participants) | 103 | 114
percentage of glycated hemoglobin | 6.9 (0.1) | 6.4 (0.1)

2. Secondary Outcome: Treatment Failure
Description: Number of participants with HbA1c>6.5% at 3 years
Time Frame: 3 years
Measure: Number; unit: number of participants
Arm/Group | Triple Therapy | Conventional Therapy
Number analyzed (Participants) | 103 | 114
number of participants | 33 | 59

3. Secondary Outcome: Percentage of Patients With Reported Hypoglycemic Events
Description: asymptomatic hypoglycemic events with documented PGC < 60 mg/dl and sympotomatic hypoglycemia
Time Frame: during the entire study (3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Triple Therapy | Conventional Therapy
Number analyzed (Participants) | 103 | 114
Participants | 14 | 52

ADVERSE EVENTS:
Time Frame: Adverse events were reported from baseline to study end (3 years) for each participant
Arm/Group | Triple Therapy | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/103 | 2/114
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/114
Other Adverse Events (participants affected / at risk) | 44/103 | 53/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple Therapy (N=103) | Conventional Therapy (N=114)
Hypoglycemia (Metabolism and nutrition disorders) | 14 (14) | 52 (52)
Nausea (Gastrointestinal disorders) | 26 (27) | 0 (0)
Peripheral Edema (Blood and lymphatic system disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT01107717/Prot_SAP_000.pdf